CLINICAL TRIAL: NCT02300220
Title: Targeted Retreatment of Incompletely Recovered COPD Exacerbations With Ciprofloxacin: a Double-blind, Randomised, Placebo-controlled, Multicentre Phase III Trial
Brief Title: Targeted Retreatment of COPD Exacerbations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14IC2031; 2012-002198-72 (EudraCT Number)
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Results first posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofloxacin (Active Comparator): 500 mg, twice daily for 1 week (oral).
  Interventions: Drug: Ciprofloxacin
- Placebo (Placebo Comparator): one capsule, twice daily for 1 week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin — 500 mg, twice daily for 1 week (oral)
  Arms: Ciprofloxacin
Drug: Placebo — One capsule, twice daily for 1 week
  Arms: Placebo

SUMMARY:
This study investigates the effects of targeted re-treatment of patients who do not recover from an exacerbation of COPD. Half of the patients will receive ciprofloxacin while the other half will receive a placebo.

DETAILED DESCRIPTION:
COPD is a long term lung condition where patients suffer recurrent symptom flare-ups, called 'exacerbations'. Patients who have lots of exacerbations have a worse quality of life, poorer ability to breath, and may die earlier than those who don't. Previous research by our group has shown that patients who have an exacerbation and have not completely recovered two weeks after the start of treatment are more likely to suffer another one early than those who completely recover.

This study aims to test whether we can prevent this early re-exacerbation by giving an extra course of antibiotics, compared to a placebo. Patients who experience an exacerbation of COPD and are treated with antibiotics will, two weeks after the start of their treatment, be invited to attend a screening visit. Patients will be eligible for the study if they have not fully recovered at this visit (i.e. if they either still have symptoms or if blood tests show there is still inflammation present) and fulfil other diagnostic measures for COPD. Patients will be allocated to the treatment groups at random, and if eligible will be treated with a further 1 week of ciprofloxacin 500mg twice daily or a placebo.

Patients will then be followed up in the study for a further 3 months, and the primary study outcome will be the time to the next exacerbation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of COPD confirmed spirometrically at screening
2. COPD exacerbation with treatment commenced 14 days prior to study enrolment and treated with 5-14 days of a non-quinolone antibiotic.
3. Exacerbation here will be defined as an episode of symptomatic worsening of COPD that was treated by the patient's attending clinician. Confirmation of the initial exacerbation diagnosis will be provided from the case notes, referral letter, or directly from the treating clinician, and will be documented in the CRF.
4. Age: ≥ 45 years of age at screening.
5. Persistent symptoms and/or a CRP≥8mg/L when assessed 2 weeks after exacerbation onset
6. Able to complete questionnaires for health status and symptoms and keep written diary cards
7. Severity of disease: Patients with a measured FEV1<80% of predicted normal values at 2 weeks post exacerbation
8. Able and willing to give signed and dated written informed consent to participate.

Exclusion Criteria:

1. Other clinically predominant chronic respiratory disease.
2. Intubated and receiving mechanical ventilation
3. Patients with known hypersensitivity to the antibiotic under evaluation, to other quinolones or any excipients of the IMP/placebo.
4. Patients with a prior history of tendonopathy or tendon rupture
5. Elderly patients taking long term systemic corticosteroids
6. Patients on long term antibiotics for other conditions
7. Patient too unwell for randomisation, i.e. requiring retreatment in the judgment of the study doctor
8. Female patients who are pregnant or planning on becoming pregnant during the study, or are breastfeeding.
9. Patient taking clinically significant contraindicated medication as per the SmPC s, such as use of concomitant tizanidine or methotrexate.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wisia Wedzicha, Professor, Principal Investigator — Imperial College London
Locations (4):
- United Kingdom (4):
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - St Georges University Hospitals NHS Foundation Trust, London
  - Royal Brompton and Harefield Hospital NHS Foundation Trust, London
  - St Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ritchie AI, Brill SE, Vlies BH, Finney LJ, Allinson JP, Alves-Moreira L, Wiseman DJ, Walker PP, Baker E, Elkin SL, Mallia P, Law M, Donaldson GC, Calverley PMA, Wedzicha JA. Targeted Retreatment of Incompletely Recovered Chronic Obstructive Pulmonary Disease Exacerbations with Ciprofloxacin. A Double-Blind, Randomized, Placebo-controlled, Multicenter, Phase III Clinical Trial. Am J Respir Crit Care Med. 2020 Aug 15;202(4):549-557. doi: 10.1164/rccm.201910-2058OC. PMID 32267724

RESULTS

PARTICIPANT FLOW:
Groups:
- Ciproflaxacin: Retreatment with Ciproflaxacin
- Placebo: Retreatment with Placebo
Period: Overall Study
Arm/Group | Ciproflaxacin | Placebo
Started | 72 | 72
Completed | 68 | 65
Not Completed | 4 | 7
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 1 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Did not tolerate IMP | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin | Placebo | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 20 | 37
  >=65 years | 55 | 52 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (8.8) | 69.1 (7.4) | 69.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 44 | 47 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 69 | 69 | 138
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 72 | 72 | 144

OUTCOME MEASURES:

1. Primary Outcome: Time to the Next COPD Exacerbation
Description: The primary outcome will be the time to the next COPD exacerbation following targeted retreatment with the IMP or placebo, censored at 90 days.
Time Frame: Up to 90 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 72 | 72
days | 72 [29 to 90] | 58 [24.5 to 90]
Statistical Analysis 1: Comparison: Ciprofloxacin vs Placebo; The primary endpoint was assessed using a Cox's proportional hazard model with pre-specified adjustment for patient's self-reported history of exacerbations over the previous year and with stratification for study centre. The onset of exacerbation will be monitored up to 90 days or at patient withdrawal; Test type: Superiority; p = 0.764, Regression, Cox; Cox Proportional Hazard = 1.071, 95% CI 2-sided [0.684 to 1.676]

2. Secondary Outcome: Duration of the Initial Exacerbation
Description: Secondary endpoints will include duration of the initial exacerbation following targeted retreatment with the IMP or placebo.
Time Frame: Up to 90 days
Population: Missing participants data 16 for ciprofloxacin and 15 for placebo
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 56 | 57
days | 3 [0 to 8] | 4 [0 to 9]
Statistical Analysis 1: Comparison: Ciprofloxacin vs Placebo; Test type: Superiority; p = 0.703, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Participants With Serious Non Fatal Adverse Events
Description: Secondary endpoints will include adverse events following targeted retreatment with the IMP or placebo.
Time Frame: 7 days of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 72 | 72
Participants | 1 | 9

4. Secondary Outcome: Changes in Lung Function
Description: Secondary endpoints will include changes from randomization to 90 days in FEV1.
Time Frame: Baseline and 90 days
Population: Only the participants who completed the study
Measure: Mean (Standard Deviation); unit: litres
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 63 | 63
litres | 0.0229 (0.199) | 0.0041 (0.198)
Statistical Analysis 1: Comparison: Ciprofloxacin vs Placebo; Test type: Superiority; p = 0.239, t-test, 2 sided

5. Secondary Outcome: Number of Participants Who Have Resistance Bacteria in the Sputum
Description: Bacterial load and resistance Secondary endpoints will include resistance following targeted retreatment with the IMP or placebo.
Time Frame: Up to 90 days
Population: Lower participants number due to the number of patients with a pathogenic organism with newly acquired ciprofloxacin resistance, present in a sputum sample collected at 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 16 | 17
Participants | 0 | 1

6. Secondary Outcome: Hospital Readmission
Description: Secondary endpoints will include hospital readmission following targeted retreatment with the IMP or placebo.
Time Frame: 90 days of treatment
Population: Data not collected
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days + 1 month
Arm/Group | Ciprofloxacin | Placebo
All-Cause Mortality (participants affected / at risk) | 1/72 | 1/72
Serious Adverse Events (participants affected / at risk) | 1/72 | 9/72
Other Adverse Events (participants affected / at risk) | 12/72 | 8/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciprofloxacin (N=72) | Placebo (N=72)
Oncology (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cardiovascular (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Psychological (Psychiatric disorders) | 0 (0) | 1 (1)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciprofloxacin (N=72) | Placebo (N=72)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Colic/Pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Pruritis/Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry Mouth (Nervous system disorders) | 1 (1) | 0 (0)
Ankle Pain/Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-07-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT02300220/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT02300220/SAP_001.pdf